CLINICAL TRIAL: NCT03665064
Title: Long Term Outcome Study in Patients With Pituitary Disorders
Status: Active, not recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00048323
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Pituitary Diseases; Pituitary Neoplasms
Keywords: Pituitary tumor; Acromegaly; Cushing; Prolactinoma
MeSH Terms: conditions — Pituitary Diseases; Pituitary Neoplasms; Acromegaly; Prolactinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the outcomes of patients with different pituitary disorders whether they are managed medically, surgically or expectantly.

DETAILED DESCRIPTION:
A chart audit of around 1500 patients seen in two specific clinics, the Medical Pituitary Clinic and the combined Endocrine/Neurosurgical Pituitary Clinic at the University of Alberta Hospital, will be performed to determine the effectiveness of various treatment strategies on the long term outcome of specific pituitary disorders. The investigator's will collect retrospective demographic (age, sex, ethnicity), clinical (mode of presentation, hormonal parameters) and therapeutic outcome (surgical, medical, expectant and / or radiation treatment; co-morbidities and complications) of patients seen in these two clinics between January 2000 and December 2020.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed pituitary disease

Exclusion Criteria:

* patients who do not have confirmed pituitary disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: tertiary referral center
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival after pituitary surgery | up to 17 years post surgery
  Using clinical, biochemical and imaging studies of a cohort of surgically operated patients to identify prognostic factors of tumor recurrence

IPD SHARING:
Plan to Share IPD: No